CLINICAL TRIAL: NCT06870786
Title: Effect of Vitamin D Deficiency on the Structure of Titanium Platelet-Rich Fibrin(T-Prf)
Brief Title: Effect of Vitamin D Deficiency on the Structure of Titanium Platelet-Rich Fibrin
Acronym: T-Prf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Esra ATEŞ, Assistan professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AibuIBU
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: PRF; Vitamin D Deficiency; Vitamin Deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Avitaminosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with vitamin D deficiency (Experimental): To obtain T-PRF membranes, blood was taken from people diagnosed with vitamin D deficiency. After 3 months, blood was taken from individuals taking vitamin D again to obtain T-PRF membranes.
  Interventions: Dietary Supplement: Vitamin D (Cholecalciferol )
- Vitamin D level is optimal (No Intervention): Blood was taken from individuals with optimum vitamin D levels to obtain T-PRF membranes

INTERVENTIONS:
Dietary Supplement: Vitamin D (Cholecalciferol ) — Evaluation of T-PRF membrane structures obtained from the blood of patients before and after vitamin D supplementation.
  Arms: with vitamin D deficiency

SUMMARY:
ABSTRACT The aim of the study was to compare the macroscopic properties, chemical degradation levels, and fibrin network structures of T-PRF membranes obtained from systemically healthy individuals with optimal vitamin D levels, with vitamin D-deficient individuals who reached optimal levels after three months of vitamin D supplementation.

A total of 48 participants, 24 with vitamin D deficiency and 24 with optimal vitamin D levels, were included in the study. The macroscopic properties (weight, width, length, density), chemical degradation levels and fibrin network structures of the obtained T-PRF membranes were evaluated using scanning electron microscopy (SEM) and light microscopy.

DETAILED DESCRIPTION:
Blood samples taken from individuals with the help of a 20 ml syringe were immediately transferred to 2 10 ml titanium tubes and placed opposite each other to ensure balance in the tabletop centrifuge device in order to be properly separated in the centrifuge process. To obtain T-PRF, it was centrifuged in the IntraSpin™ device at 2700 rpm centrifugal force for 12 minutes.

After centrifugation, the fibrin in the middle of the 3 layers formed in the titanium tube was held and pulled with the help of a press. Then, the red layer in the lower layer, where erythrocytes were dense, was separated from the fibrin layer with the help of scissors and the membrane was obtained by pressing for 2 minutes using the own weight of the PRF box.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20-55
* Being systemically healthy
* Not using any medication regularly
* Not taking additional vitamin D from outside
* Patients who met the conditions of not having used antibiotics for the last three months were included in the study.

Exclusion Criteria:

* People who use cigarettes (tobacco) and alcohol
* Those with platelet function and clotting disorders
* Those who are pregnant or breastfeeding
* Those who use medications that affect the natural clotting process
* Those with a history of infection in the last three months
* Those receiving immunosuppressive therapy
* Those who do not consent to volunteer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
microscopic analysis | From enrollment to the end of treatment at 3 months
  T-PRF membranes were examined histologically using the cell block cytology method. Membranes were transferred to cassettes and fixed in formalin solution for 24 hours. At the end of 24 hours, the cassettes were subjected to dehydration with various concentrations of formalin, alcohol and xylene. The tissue was embedded in Leucher blocks using paraffin so that it could be easily cut and examined. 3 µm thick sections were taken from the embedded blocks using a microtome. Paraffin in the blocks was removed and the tissue was stained with hematoxylin-eosin L-PRF clot was analyzed microscopically on hematoxylin-eosin stained slides using the blood element adhesion index score 0: absence of fibrin network score 1: sparsely dispersed fibrin network score 2: thin fibrin network poorly interlocking score 3: dense fibrin network abundantly interconnected

SECONDARY OUTCOMES:
Scanning Electron Microscope (SEM) Examination | From enrollment to the end of treatment at 3 months
  In order to visualize the surfaces of the samples, they were coated with 20 nm gold/palladium sputtering and photographs were taken and recorded under different magnifications.
T-PRF Degradation of Membranes | From enrollment to the end of treatment at 3 months
  T-PRF membranes weighed was placed in an orbital shaking device in 7.4% PBS solution for 1 week in order to evaluate the degradation rates Degradation amounts were calculated as:% degradation=(initial weight-final weight)/initial weight x 100

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Bolu Abant İzzet Baysal University,, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No